CLINICAL TRIAL: NCT05471271
Title: An Open Label Pilot Study of [18AlF]-RESCA-IL2 (Interleukin-2 PET Tracer) for Positron Emission Tomography Imaging in Patients Treated With Immune Checkpoint Inhibitors.
Brief Title: IL-2 PET Imaging in Advanced Solid Tumours
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Instability of the IL2 tracer
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202100912
Record Dates: First submitted 2022-06-29; First posted 2022-07-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18AlF]-RESCA-IL2 PET imaging (Other)
  Interventions: Other: [18F]AlF-RESCA-IL2 PET scan

INTERVENTIONS:
Other: [18F]AlF-RESCA-IL2 PET scan — Patients will undergo [18F]AlF-RESCA-IL2 PET imaging twice; the first [18F]AlF-RESCA-IL2 PET scan will be performed at baseline, before starting therapy. The second [18F]AlF-RESCA-IL2 PET scan will be performed after 2 weeks of treatment

SUMMARY:
This is an investigator-initiated, single-center, open-label clinical trial designed to evaluate the safety and PK of the PET tracer [18F]AlF-RESCA-IL2 in patients prior to and during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing informed consent.
2. Patients with histologically confirmed diagnosis of locally advanced or metastatic solid cancer, eligible for ICI therapy as part of routine care.
3. At least 1 lesion that is accessible per investigator's assessment and eligible for biopsy according to standard clinical care procedures.
4. Measurable disease, as defined by standard RECIST v1.1. Previously irradiated lesions should not be counted as target lesions except for lesions that have progressed after radiotherapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy ≥ 12 weeks.
7. Signed informed consent.
8. Willingness and ability to comply with all protocol required procedures.
9. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception (i.e., one that results in a low failure rate (< 1% per year) when used consistently and correctly)).

Exclusion Criteria:

1. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to [18F]AlF-RESCA-IL2 injection.
2. Evidence of an active infection that requires systemic antibiotics within 2 weeks prior to [18F]AlF-RESCA-IL2 injection.
3. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of [18F]AlF-RESCA-IL2, or that may affect the interpretation of the results or render the patient at high risk from complications.
4. Altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
5. Sponsor employee/member of the clinical site study team and/or his or her immediate family
6. Pregnant or lactating females.
7. Concurrent use of systemic corticosteroids > 10 mg daily prednisone equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events related to [18F]-AlF-RESCA-IL2 administration as assessed by CTCAE v5.0 | 2 years
  Safety assessment through summaries of adverse events, changes in laboratory test results (if evaluation is indicated) and changes in vital signs. Adverse event data will be recorded and summarized according to NCI CTCAE v5.0
Non-displaceable binding potential (BPND) | 2 years
  To evaluate the pharmacokinetic behaviour of 18F-AIF-RESCA-IL2 through activity in venous blood samples, dynamic imaging, and pharmacokinetic modeling.
Total volume of distribution (VT) of the tracer in the tumour | 2 years
  To evaluate the pharmacokinetic behaviour of 18F-AIF-RESCA-IL2 through activity in venous blood samples, dynamic imaging, and pharmacokinetic modeling.
Biodistribution of [18F]-AlF-RESCA-IL2 | 2 years
  Evaluation of [18F]AlF-RESCA-IL2 biodistribution in cancer patients on the PET images by measuring standardized uptake values in tumours, healthy tissues and organs.

SECONDARY OUTCOMES:
Correlation of 18F-AlF-RESCA-IL2 uptake in tumours, with T cell infiltration in tumour biopsy samples, as determined by IHC. | 2 years
  Results of immunohistochemical (IHC) scoring of immune cell IL-2R expression will be described as a semi-quantitative score using the percentage of positive cells (continuous variable), intensity and pattern of staining (discrete variable). These IHC results will be compared with imaging tracer standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the PET scan images.
Correlation of 18F-AlF-RESCA-IL2 PET measurements with radiologic response to treatment, according to (i)RECIST v1.1 criteria. | 2 years
  Response to therapy will be assessed according to the RECIST or iRECIST guidelines. These results will be compared with imaging tracer standardized uptake value (SUV) in defined volumes of interest (VOIs) of tumor lesions on the PET scan images.
Assessment of changes in tumour and normal organ tracer uptake after 2 weeks of treatment, expressed as standardized uptake values. | 2 years
  Patients will undergo a PET scan at baseline and another one during treatment. tracer uptake will be quantified and expressed as standardized uptake value (SUV) in defined volumes of interest (VOIs) for both scans. The results of both PET scans will be compared to assess changes in imaging tracer uptake over time.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No